CLINICAL TRIAL: NCT01033123
Title: A Phase 2, Multi-Center, Single-Arm Study Evaluating Carboplatin/Gemcitabine in Combination With BSI-201 in Patients With Platinum-Sensitive Recurrent Ovarian Cancer
Brief Title: A Single-Arm Study Evaluating Carboplatin/Gemcitabine in Combination With BSI-201 in Patients With Platinum-Sensitive Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11503; 20090207 (Other: BiPar)
Expanded Access: NCT01130259 (No longer available)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian; cancer; sensitive; PARP; recurrent; platinum-sensitive recurrent ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Hypersensitivity; Recurrence | interventions — iniparib; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BSI-201 (Experimental): BSI-201 in combination with gemcitabine and carboplatin.
  Interventions: Drug: BSI-201

INTERVENTIONS:
Drug: BSI-201 — IV infusion, 5.6 mg/kg
  Other Names: PARP inhibitor

SUMMARY:
The purpose of this study is to evaluate the effect of BSI-201 on the objective response rate in platinum-sensitive recurrent ovarian cancer patients receiving gemcitabine and carboplatin.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histological diagnosis of epithelial ovarian carcinoma, fallopian tube cancer, or primary peritoneal carcinoma
* Completion of only one previous course of chemotherapy which contained a platinum therapy, with sensitivity to that regimen. "Platinum-sensitivity" is defined by a relapse greater than 6 months after termination of platinum-based chemotherapy
* Measurable disease, defined by at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded), and is ≥ 20 mm when measured by conventional techniques (palpation, plain x-ray, computed tomography [CT], or magnetic resonance imaging [MRI]) or ≥ 10 mm when measured by spiral CT
* Adequate organ function defined as: absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3, creatinine clearance > 50mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN; or < 5 x ULN in case of liver metastases); total bilirubin < 1.5 mg/dL
* For women of child bearing potential, documented negative pregnancy test within two weeks of study entry and agreement to acceptable birth control during the duration of the study therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Signed, institutional review board (IRB) approved written informed consent

Exclusion Criteria:

* Concurrent invasive malignancy, not including:

  1. Non-melanomatous skin cancer
  2. In situ malignancies
  3. Concurrent superficial endometrial carcinoma, if their endometrial carcinoma is superficial or invades less than 50% the thickness of the myometrium)
  4. Low risk breast cancer (localized, non-inflammatory) treated with curative intent
* Lesions identifiable only by positron emission tomography (PET)
* Prior treatment with poly (ADP-ribose) polymerase (PARP) inhibitors, including BSI-201
* Major medical conditions that might affect study participation (i.e., uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection)
* Other significant co-morbid condition which the investigator feels might compromise effective and safe participation in the study, including a history of congestive cardiac failure or an electrocardiogram (ECG) suggesting significant conduction defect or myocardial ischemia
* Enrollment in another investigational device or drug study, or current treatment with other investigational agents
* Concurrent radiation therapy to treat primary disease throughout the course of the study
* Inability to comply with the requirements of the study
* Pregnancy or lactation
* Leptomeningeal disease or brain metastases requiring steroids or other therapeutic intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the objective response rate (ORR) of gemcitabine/carboplatin in combination with BSI-201 | Until progressive disease or death

SECONDARY OUTCOMES:
To determine the nature and degree of toxicity of gemcitabine/carboplatin in combination with BSI-201 | 30 days after last BSI-201 exposure
To evaluate progression-free survival (PFS) of gemcitabine/carboplatin in combination with BSI-201 | until progressive disease or death

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Massachusetts Ceneral Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Penson RT, Ambrosio AJ, Whalen CA, Krasner CN, Konstantinopoulos PA, Bradley C, Matulonis UA, Birrer MJ. Phase II Trials of Iniparib (BSI-201) in Combination with Gemcitabine and Carboplatin in Patients with Recurrent Ovarian Cancer. Oncologist. 2023 Mar 17;28(3):252-257. doi: 10.1093/oncolo/oyac275. PMID 36718018